CLINICAL TRIAL: NCT03278821
Title: A Randomized Controlled Study of Patients Matching Themselves to Treatment Options: The Self-Match Study
Brief Title: The Self Match Study: A Study of Informed Choice in the Treatment of Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kjeld Andersen (Other)
Responsible Party: Sponsor-Investigator, Kjeld Andersen, Professor, University of Southern Denmark
Organization: University of Southern Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RESCueH, The Self Match Study
Record Dates: First submitted 2017-03-29; First posted 2017-09-12 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Alcohol Dependence
Keywords: Informed choice; Alcohol use disorder; Addiction treatment
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self Match (Experimental): The patient must choose between the five possible treatment options.
  Interventions: Behavioral: Self Match
- Expert Match (Active Comparator): The Patient is referred to treatment by standard procedure which is Expert Match based on patient data.
  Interventions: Behavioral: Expert Match

INTERVENTIONS:
Behavioral: Self Match — Video presentation of treatment option are shown to the patient whereafter the patient must choose between the five possible treatment options.
  Arms: Self Match
Behavioral: Expert Match — Referral as usual to one of five possible treatment options. The referral is based on baseline data from the patient and by the means of an algorithm, used in daily clinical praxis.
  Arms: Expert Match

SUMMARY:
The purpose of this study is to determine whether patient self-matching (as compared with treatment as usual by expert matching) improves quality of life, retention, and outcome for patients being treated for alcohol problems.

There are at least two good reasons for offering patients a choice when the goal is a change in their behavior. The first is that patients are likely to know what treatment works best for them. Secondly, being allowed to choose between options may increase compliance in treatment. As a randomized controlled trial, this study will compare the efficacy of patient self-matching versus treatment-as-usual expert matching.

The Self-Match Study is expected to increase knowledge on the importance of involving the alcohol dependent patient in choosing what treatment method is best for him/her instead of having experts to do that. The investigators expect to discover patient involvement as a way to improve compliance in treatment, hence preventing that patients drop out of treatment to early. If this hypothesis proves to be right, clinicians will have a viable strategy for matching treatment methods to patients, since the strategy does not demand further resources in the treatment system.

ELIGIBILITY:
Inclusion Criteria:

1. Fulfilling DSM-IV criteria for alcohol abuse or dependence.
2. Native Danish speaking.
3. Having no severe psychosis or cognitive impairment.
4. Accepting to participate in the study.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
Reduced amount of drinking days measured by Time Line Follow Back. | 6 months after initiation of treatment.
  The primary endpoint analysis will be a comparison of outcomes for patients assigned to the self-match group vs. expert-match group to determine whether self-matching yields more favorable outcome than expert matching, measured by the number of excessive drinking days.

SECONDARY OUTCOMES:
Compliance measured by proportion of patients who has completed treatment. | 6 months after treatment start
  Data on patients who have completed treatment as planned will be gathered from treatment journal.
Quality of life measured by WHO's Quality of Life scale. | 6 months after treatment start.
  Patients reporting increase or decrease in quality of life compared to baseline.
Personality traits, measured by NEO-FFI-3, influence on outcome. | 6 months after treatment start.
  Comparison of personality traits with outcome measures.
Deviation in the chosen treatment in the Self-Match group in relation to the expected expert choice. | 6 months after treatment start.
  The algorithm score used in expert-matching will be calculated for all patients. The chosen treatment for patients in The Self-Match Group will be compared to the algorithm score to measure convergence between Self-Match and Expert-Match.

CONTACTS AND LOCATIONS:
Locations (1):
- RESCueH alcohol Studies, Unit of Clinical Alcohol Research, Psyciatric Research Unit, Clinical Institute, University of Southern Denmark, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hell ME, Miller WR, Nielsen B, Nielsen AS. Is treatment outcome improved if patients match themselves to treatment options? Study protocol for a randomized controlled trial. Trials. 2018 Apr 6;19(1):219. doi: 10.1186/s13063-018-2592-9. PMID 29625579

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT03278821/SAP_000.pdf